CLINICAL TRIAL: NCT04725357
Title: A Randomized Comparison of Meloxicam to Opioids Following Arthroscopic Labrum Repairs of the Shoulder
Brief Title: Does Meloxicam Provide as Much Pain Relief as Opioids After Shoulder Surgery?
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JHOR20D.1216
Record Dates: First submitted 2021-01-18; First posted 2021-01-26 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Meloxicam

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arthroscopic Labral Repair + postoperative Meloxicam (Experimental): After surgery participants will receive a prescription of 20 pills of 15 mg Meloxicam
  Interventions: Drug: Meloxicam 15 mg; Procedure: Preoperative Interscalene Nerve Block; Procedure: arthroscopic labral repair
- Arthroscopic Labral Repair without Meloxicam (Active Comparator): After surgery participants will receive a prescription of 20 pills of 5/300 mg vicodin (hydrocodone/acetaminophen)
  Interventions: Procedure: Preoperative Interscalene Nerve Block; Procedure: arthroscopic labral repair

INTERVENTIONS:
Drug: Meloxicam 15 mg — Participants will receive a prescription of 20 pills of 15 mg Meloxicam after surgery
  Arms: Arthroscopic Labral Repair + postoperative Meloxicam
Procedure: Preoperative Interscalene Nerve Block — Preoperatively participants will standardly receive an interscalene nerve block
Procedure: arthroscopic labral repair — participant will have their standard surgical procedure done

SUMMARY:
The opioid epidemic continues to be a major concern, with orthopedic surgeons being among the top prescribers of opioids. Studies evaluating these practices found that opioids are overprescribed, even for common procedures. Patients undergoing arthroscopic labrum repair of the shoulder were found to have an average of 20 pills left over after surgery. Many strategies have been developed to tackle overprescribing and have found success, including no opioid protocols for carpal tunnel release. The purpose of this study is to examine if meloxicam alone provides similar patient reported outcomes to opioids following arthroscopic labrum repair of the shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18
* Scheduled for arthroscopic labrum repair of the shoulder

Exclusion Criteria:

* History of opioid, acetaminophen, NSAID or local anesthetic allergy or intolerance, or contraindications to these medications.
* Currently on long-term preoperative narcotics
* Scheduled for revision arthroscopic repairs of the shoulder
* Unable/unwilling to consent for enrollment
* Unable to complete postoperative surveys
* History of chronic pain syndromes (fibromyalgia, chronic diffuse MSK pain, etc)
* Patients under the age of 18
* Pregnant or breastfeeding women
* Scheduled for concurrent procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-01-25 (Estimated); Primary Completion 2022-01-25 (Estimated); Study Completion 2022-01-25 (Estimated)

PRIMARY OUTCOMES:
Total Analgesic use | 14 days
  Participants will be given a survey asking about number of pills taken
Postoperative Pain Control | 14 days
  Measured by the Numerical Rating Scale (NRS) pain score daily after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Philadelphia, Pennsylvania, United States